CLINICAL TRIAL: NCT05825755
Title: Randomized Controlled Multicenter Trial for the Validation of Vitalera Platform
Brief Title: Multicenter Trial for the Validation of Vitalera Platform
Acronym: VAL-HIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: humanITcare (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FOLLOWHEALTH-2023-02
Record Dates: First submitted 2023-03-24; First posted 2023-04-24 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Chronic Patients; Heart Failure
Keywords: Chronic care; Chronic patients; Heart Failure; Telemonitoring; Remote monitoring; Remote care; Healthcare; Home care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (UC) (No Intervention): The follow-up of the patients in the UC arm will be carried out in accordance with the usual clinical practice of each recruitment center. All recruiting centers have active and mature HF programs in place and therefore each center will decide how to follow up the patient. However, medical professionals will be required to register each patient on the platform, enter their baseline data (sociodemographics and risk factors) and enter all possible clinical events (death, non-fatal HF event, hospitalization or emergency room visit). that the patient could suffer during the entire follow-up period.
  The number of pre-planned contacts will be defined according to the particular clinical practice of each recruitment center.
- Telemonitoring (TM) (Experimental): Patients in the TM arm will be followed up with the vitalera platform and app. Physiological parameters (measured periodically), socio-demographic data, risk factors, medication tracking, symptomatology questionnaire for patients, NYHA-class, clinical interventions, health questionnaire answers, classified alarms with their respective timestamp and annotation by the MD, and measurement ranges for each personalized alarm and their changes.
  Interventions: Other: vitalera telemonitoring platform

INTERVENTIONS:
Other: vitalera telemonitoring platform — Patients will be followed-up with measurements from medical devices and health questionnaires delivered through the app
  Arms: Telemonitoring (TM)

SUMMARY:
Vitalera has implemented a cloud platform for the telemonitoring of chronic patients through portable medical devices and an alarm-based system that issues health alerts when a patient's biomedical measurement is outside a predefined clinical range. The platform frees doctors and caregivers from reviewing individual patient data for abnormalities, speeding up the decision-making process and reducing hospital visits. With this study we intend to validate the efficacy of the app for patients and digital platform for medical professionals, evaluating the increase in the quality of life of patients and measuring the reduction in the incidence of the main critical events of HF. In addition, the study will validate the new API interoperability standards and platform architecture and will assess the usability of the platform by delivering satisfaction questionnaires to patients and professionals at the end of the study.

This study is being carried out within the framework of a European project promoted by the European Innovation Council (EIC).

DETAILED DESCRIPTION:
This is a randomized controlled trial involving a Spanish network of hospitals. The study consists of continuous remote patient monitoring using vitalera's digital platform and the supplied devices (blood pressure monitor, wearable, scale and oximeter). For 3 months, a total of 250 patients suffering from HF will have their physiological constants monitored.

Patients will be included in the study based on the eligibility criteria and must complete the informed consent provided. Each hospital will decide when to include their patients according to their particular clinical practice. The recruitment period is defined as 3 months. That means patients will be incorporated into the study from its start until the third month. The last subject included in the study will then finish the study after six months from the first day of the study. Medical professionals from each hospital will be in charge of recruiting the participants. The recruitment rate is specific for each hospital, and it may vary depending on the month.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure (HF) patients with NYHA Functional Class >= II (according to 2021 EU guidelines).
* Patients older than 18 years old.
* Patients who have suffered an acute decompensation of HF (first and recurrent) in the 30 days prior to enrollment in the study.
* NT-pro BNP ≥300 pg/ml at the moment of hospitalization for patients without ongoing atrial fibrillation/flutter. If ongoing atrial fibrillation/flutter, NT-pro BNP must be ≥600 pg/mL
* Patients must have had an echocardiogram during their HF hospitalization or in the previous 12 months.
* Prior to initiating any procedures, the hospital will ensure that the patient obtains an informed consent document, if applicable.
* All patients will be eligible regardless of the level of LVEF: HFrEF, HFmrEF, and HFpEF.

Exclusion Criteria:

* Oncology patients with metastasis or with chemotherapy treatment ongoing
* Patients participating in other studies or trials.
* Patients not willing to participate.
* Patients over 150 kg
* Patients who do not use Catalan, Spanish, English, Portuguese, Italian, Dutch, German, Swedish, Hungarian, Romanian or French.
* Patients without a mobile phone
* Patients without internet connexion
* Patients with moderate or severe cognitive impairment without a competent caregiver
* Patients with serious psychiatric illness
* Patients with planned cardiac surgery
* Patients with planned heart transplantation or LVAD implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta MD Farrero, Principal Investigator — Hospital Clinic of Barcelona
Locations (10):
- Spain (10):
  - Hospital de Dénia, Denia, Alacant
  - Hospital d'Alcoi, Alcoy, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital de Vinalopó, Elche, Alicante
  - Hospital de Terrassa, Terrassa, Barcelona
  - Corporació de Salut del Maresme i la Selva (Hospital de Blanes-Hospital de Calella), Blanes, Girona
  - Hospital de Torrejón, Torrejón de Ardoz, Madrid
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Clínico Lozano Blesa de Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tripoliti EE, Papadopoulos TG, Karanasiou GS, Naka KK, Fotiadis DI. Heart Failure: Diagnosis, Severity Estimation and Prediction of Adverse Events Through Machine Learning Techniques. Comput Struct Biotechnol J. 2016 Nov 17;15:26-47. doi: 10.1016/j.csbj.2016.11.001. eCollection 2017. PMID 27942354
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2022 Jan;24(1):4-131. doi: 10.1002/ejhf.2333. PMID 35083827
- [Background] Schiff GD, Fung S, Speroff T, McNutt RA. Decompensated heart failure: symptoms, patterns of onset, and contributing factors. Am J Med. 2003 Jun 1;114(8):625-30. doi: 10.1016/s0002-9343(03)00132-3. PMID 12798449
- [Background] Brahmbhatt DH, Cowie MR. Remote Management of Heart Failure: An Overview of Telemonitoring Technologies. Card Fail Rev. 2019 May 24;5(2):86-92. doi: 10.15420/cfr.2019.5.3. eCollection 2019 May. PMID 31179018
- [Background] Scherr D, Kastner P, Kollmann A, Hallas A, Auer J, Krappinger H, Schuchlenz H, Stark G, Grander W, Jakl G, Schreier G, Fruhwald FM; MOBITEL Investigators. Effect of home-based telemonitoring using mobile phone technology on the outcome of heart failure patients after an episode of acute decompensation: randomized controlled trial. J Med Internet Res. 2009 Aug 17;11(3):e34. doi: 10.2196/jmir.1252. PMID 19687005
- [Background] Koulaouzidis G, Iakovidis DK, Clark AL. Telemonitoring predicts in advance heart failure admissions. Int J Cardiol. 2016 Aug 1;216:78-84. doi: 10.1016/j.ijcard.2016.04.149. Epub 2016 Apr 21. PMID 27140340
- [Background] Koehler F, Winkler S, Schieber M, Sechtem U, Stangl K, Bohm M, Boll H, Baumann G, Honold M, Koehler K, Gelbrich G, Kirwan BA, Anker SD; Telemedical Interventional Monitoring in Heart Failure Investigators. Impact of remote telemedical management on mortality and hospitalizations in ambulatory patients with chronic heart failure: the telemedical interventional monitoring in heart failure study. Circulation. 2011 May 3;123(17):1873-80. doi: 10.1161/CIRCULATIONAHA.111.018473. Epub 2011 Mar 28. PMID 21444883
- [Background] Lee S, Chu Y, Ryu J, Park YJ, Yang S, Koh SB. Artificial Intelligence for Detection of Cardiovascular-Related Diseases from Wearable Devices: A Systematic Review and Meta-Analysis. Yonsei Med J. 2022 Jan;63(Suppl):S93-S107. doi: 10.3349/ymj.2022.63.S93. PMID 35040610
- [Background] Guidi G, Pollonini L, Dacso CC, Iadanza E. A multi-layer monitoring system for clinical management of Congestive Heart Failure. BMC Med Inform Decis Mak. 2015;15 Suppl 3(Suppl 3):S5. doi: 10.1186/1472-6947-15-S3-S5. Epub 2015 Sep 4. PMID 26391638
- [Background] Jaarsma T, Arestedt KF, Martensson J, Dracup K, Stromberg A. The European Heart Failure Self-care Behaviour scale revised into a nine-item scale (EHFScB-9): a reliable and valid international instrument. Eur J Heart Fail. 2009 Jan;11(1):99-105. doi: 10.1093/eurjhf/hfn007. PMID 19147463
- [Background] Roque NA, Boot WR. A New Tool for Assessing Mobile Device Proficiency in Older Adults: The Mobile Device Proficiency Questionnaire. J Appl Gerontol. 2018 Feb;37(2):131-156. doi: 10.1177/0733464816642582. Epub 2016 Apr 11. PMID 27255686
- [Background] Bilbao A, Escobar A, Garcia-Perez L, Navarro G, Quiros R. The Minnesota living with heart failure questionnaire: comparison of different factor structures. Health Qual Life Outcomes. 2016 Feb 17;14:23. doi: 10.1186/s12955-016-0425-7. PMID 26887590

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care (UC): The follow-up of the patients in the UC arm will be carried out in accordance with the usual clinical practice of each recruitment center. All recruiting centers have active and mature HF programs in place and therefore each center will decide how to follow up the patient. However, medical professionals will be required to register each patient on the platform, enter their baseline data (sociodemographics and risk factors) and enter all possible clinical events (death, non-fatal HF event, hospitalization or emergency room visit). that the patient could suffer during the entire follow-up period. In addition, patients will use the app only to answer to health questionnaires in order to stardardize the responses from both group and evaluate the outcomes of the study.
  The number of pre-planned contacts will be defined according to the particular clinical practice of each recruitment center.
Period: Overall Study
Arm/Group | Usual Care (UC) | Telemonitoring (TM)
Started | 45 | 52
Completed | 43 | 44
Not Completed | 2 | 8

BASELINE CHARACTERISTICS:
Population: Patients that abandoned the study (10 patients) weren't considered for analysis. Those considered for all the analysis were the ones that completed plus the deseased patients (2 patients).
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care (UC) | Telemonitoring (TM) | Total
Number analyzed (Participants) | 43 | 46 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (13) | 66 (16) | 68 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 30 | 35 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 36 | 44 | 80
  Ethnicity: Latino | 6 | 2 | 8
  Ethnicity: Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Spain | 43 | 46 | 89
NYHA class [Count of Participants; unit: Participants] — The NYHA Functional Classification assesses heart failure severity based on physical activity limitations and symptoms like dyspnea, fatigue, and palpitations. It guides treatment decisions and monitors progression:
  Class I: No symptoms with ordinary activity. Class II: Slight limitation; symptoms with ordinary activity. Class III: Marked limitation; symptoms with less than ordinary activity. Class IV: Symptoms at rest or with minimal activity.
  Ref: McDonagh, et al. "2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure(...)" European Heart Journal
  Participants
    II | 28 | 22 | 50
    III | 12 | 19 | 31
    IV | 3 | 5 | 8
LVEF categorical [Count of Participants; unit: Participants] — Left Ventricular Ejection Fraction (LVEF) measures the percentage of blood the left ventricle pumps with each heartbeat, essential for heart failure (HF) classification:
  HFrEF: LVEF ≤ 40% (reduced) HFmrEF: LVEF 41-49% (mildly reduced) HFpEF: LVEF ≥ 50% (preserved) HFimpEF: Previously ≤ 40%, now > 40% with improvement LVEF guides HF diagnosis, treatment, and prognosis. McDonagh, et al. "2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure (...)" European heart journal 42.36 (2021): 3599-3726.
  Participants
    < 40 | 21 | 32 | 53
    40 - 50 | 7 | 5 | 12
    >= 50 | 15 | 9 | 24
Employment status [Count of Participants; unit: Participants]
  Retired | 26 | 28 | 54
  Paid | 13 | 14 | 27
  None | 2 | 2 | 4
  Unemployed | 0 | 2 | 2
  Voluntary work | 1 | 0 | 1
  Student | 1 | 0 | 1
Education level [Count of Participants; unit: Participants]
  Primery | 12 | 10 | 22
  Secondary | 14 | 20 | 34
  High level | 9 | 12 | 21
  No education | 8 | 4 | 12
Does the patient have caretaker? [Count of Participants; unit: Participants]
  Yes | 20 | 17 | 37
  No | 23 | 29 | 52
Number of people living with the patient [Mean (Standard Deviation); unit: people] | 2 (1) | 2 (1) | 2 (1)
Smoker [Count of Participants; unit: Participants]
  Yes | 9 | 4 | 13
  No | 15 | 20 | 35
  Ex-smoker | 19 | 22 | 41
Alcohol use [Count of Participants; unit: Participants]
  Yes | 2 | 5 | 7
  Yes, occasionally | 18 | 19 | 37
  No | 23 | 22 | 45
Diabetes [Count of Participants; unit: Participants]
  Yes | 11 | 14 | 25
  No | 32 | 32 | 64
Hypertension [Count of Participants; unit: Participants]
  Yes | 27 | 26 | 53
  No | 16 | 20 | 36
Heart disease history [Count of Participants; unit: Participants]
  Yes | 34 | 35 | 69
  No | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life Scale Between Baseline and 3-months Follow-up
Description: Quality of life measured with the Minnesota Living with Heart Failure scale. Scale from 0 to 105. The lower the score the better outcome.
Time Frame: 3 months
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care (UC) | Telemonitoring (TM)
Number analyzed (Participants) | 38 | 40
units on a scale | -24 [-24.5 to -8] | -32.5 [-33.5 to -9.5]
Statistical Analysis 1: Comparison: Usual Care (UC) vs Telemonitoring (TM); Test type: Superiority; p = 0.252, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in the Proportion of Treatment Adherent Patients Between Baseline and 3-months Follow-up.
Description: Change in the proportion of patients adherent to treatment measured with SMAQ between start and end of the study. This questionnaire consists of six questions that evaluate different aspects of patient compliance with treatment: forgetfulness, routine, adverse effects, and a quantification of omissions. A patient is classified as non-compliant (non-adherent) if he/she responds to any of the questions with a non-adherence answer, and in terms of quantification, if the patient has lost more than two doses during the last week or has not taken medication during more than two complete days during the last three months.
  Then we compute the proportion of adherent patients at baseline and 3-months follow-up and compute the change in proportion.
Time Frame: 3 months
Measure: Number; unit: proportion of participants
Arm/Group | Usual Care (UC) | Telemonitoring (TM)
Number analyzed (Participants) | 36 | 39
proportion of participants | 0.056 | 0.068
Statistical Analysis 1: Comparison: Usual Care (UC) vs Telemonitoring (TM); Test type: Superiority; p = 1.0, McNemar

3. Primary Outcome: Change in Sel-care Behaviour Scale Between Baseline and 3-months Follow-up
Description: Patient's self-care behavior measured with The European Heart Failure Self-Care Behavior Scale. Scale from 9 to 45. The higher the score the poorer self-care.
Time Frame: 3 months
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care (UC) | Telemonitoring (TM)
Number analyzed (Participants) | 39 | 39
units on a scale | -4 [-7 to 0] | -4 [-7 to -1]
Statistical Analysis 1: Comparison: Usual Care (UC) vs Telemonitoring (TM); Test type: Superiority; p = 0.791, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Mortality From Any Cause
Description: Number of deaths during the study period
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Telemonitoring (TM)
Number analyzed (Participants) | 43 | 46
Participants | 0 | 2

5. Secondary Outcome: Number of Hospital Readmissions
Description: Total number of hospitalizations
Time Frame: 3 months
Measure: Number; unit: hospitalizations
Arm/Group | Usual Care (UC) | Telemonitoring (TM)
Number analyzed (Participants) | 43 | 46
hospitalizations | 7 | 7

6. Secondary Outcome: Number of Visits to the Emergency Room Due to HF Decompensation
Description: Total number of visits with intravenous decongestive therapy
Time Frame: 3 months
Measure: Number; unit: visits to emergency room
Arm/Group | Usual Care (UC) | Telemonitoring (TM)
Number analyzed (Participants) | 43 | 46
visits to emergency room | 2 | 0

7. Secondary Outcome: Number of Emergency Visits for CV Causes
Description: Total number of visits due to cardiovascular causes
Time Frame: 3 months
Measure: Number; unit: visits to emergency room
Arm/Group | Usual Care (UC) | Telemonitoring (TM)
Number analyzed (Participants) | 43 | 46
visits to emergency room | 3 | 1

ADVERSE EVENTS:
Time Frame: During 3-month follow-up
Arm/Group | Usual Care (UC) | Telemonitoring (TM)
All-Cause Mortality (participants affected / at risk) | 0/43 | 2/46
Serious Adverse Events (participants affected / at risk) | 9/43 | 7/46
Other Adverse Events (participants affected / at risk) | 3/43 | 1/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (UC) (N=43) | Telemonitoring (TM) (N=46)
All-cause hospitalizaton (Cardiac disorders) | 7 (7) | 7 (7)
Urgent visit with intravenous decongestive therapy (Cardiac disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (UC) (N=43) | Telemonitoring (TM) (N=46)
Visit to medical emergencies (Cardiac disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT05825755/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT05825755/ICF_001.pdf